CLINICAL TRIAL: NCT01608841
Title: The Role of Epidermal Growth Factor Receptor (EGFR) Mutations in Pancreatic Cancer Patients Receiving Gemcitabine With or Without Erlotinib
Brief Title: The Role of EGFR Mutations in Pancreatic Cancer Patients Receiving Gemcitabine With or Without Erlotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Attending Physician, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 98-01-34A
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine (No Intervention)
- Gemcitabine plus erlotinib (Experimental)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 100 mg 1# PO qd till disease progression
  Other Names: Tarceva
  Arms: Gemcitabine plus erlotinib

SUMMARY:
The purpose of this study is to investigate the influence of epidermal growth factor receptor mutations on the efficacy of erlotinib and gemcitabine in metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The influence of EGFR mutations on the efficacy of treatment with and without erlotinib in metastatic pancreatic cancer is to be determined.

ELIGIBILITY:
Inclusion Criteria:

* metastatic chemotherapy-naïve pancreatic cancer patients
* histologically confirmed
* adequate samples for analysis
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2
* absolute neutrophil count (ANC) >= 1,500/mm3
* platelet count >= 100,000/mm3
* serum creatinine <= 1.5 mg/dL
* aspartate aminotransferase (AST)
* alanine aminotransferase (ALT) < 5 times the upper limit of normal

Exclusion Criteria:

* absence of any other malignancy or serious medical or psychological illness that would preclude informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2005-07; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
disease control rate | eight weeks

SECONDARY OUTCOMES:
response rate | eight weeks
overall survival | one day
progression-free survival | one day

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Pin Li, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Yee Chao, MD,PhD, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Division of Gastroenterology, Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Wang JP, Wu CY, Yeh YC, Shyr YM, Wu YY, Kuo CY, Hung YP, Chen MH, Lee WP, Luo JC, Chao Y, Li CP. Erlotinib is effective in pancreatic cancer with epidermal growth factor receptor mutations: a randomized, open-label, prospective trial. Oncotarget. 2015 Jul 20;6(20):18162-73. doi: 10.18632/oncotarget.4216. PMID 26046796